CLINICAL TRIAL: NCT04251845
Title: Evaluation of Effect of Topical Melatonin in Treatment of Oral Leukoplakia: A Randomized Placebo Controlled Study
Brief Title: Evaluation of Effect of Topical Melatonin in Treatment of Oral Leukoplakia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shubhangi OMR
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Oral Leukoplakia
MeSH Terms: conditions — Leukoplakia, Oral | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Active Comparator): Intervention : Topical Melatonin(3%) at dosage of 15 mg once daily
  Interventions: Dietary Supplement: topical melatonin
- Control Group (Placebo Comparator): Intervention : Placebo once daily
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: topical melatonin — Topical melatonin at 3% concentration with dosage of 15 mg once daily will be applied on the lesion for 6 weeks followed by a follow up of 3 months
  Arms: Trial group
Other: PLACEBO — Topical application of placebo once daily for 6 weeks with a follow up for 3 months
  Arms: Control Group

SUMMARY:
Oral leukoplakia is the most commonly occurring oral premalignant disorder. It has an overall prevalence rate of 1-4% with highest prevalence rate of 10.54% in Asian countries. The management of leukoplakia includes conventional as well as surgical modalities. The conventional approaches include Beta Carotene, Lycopene, ascorbic acid, alpha tocopherol, retinoids. But, no significant results are documented on regression rate and prevention of recurrence of the lesions.

Melatonin chemically N-acetyl-5-methoxytryptamine is a hormone produced in the pineal gland. It is synthesized from the amino acid, tryptophan. The basic physiological function of melatonin is to control day night cycle and hence is commonly used in insomnia, jet lag and some other psychological disorders.

Melatonin has a potent antioxidant effect and other actions such as modulation of cell cycle and induction of apoptosis, inhibition of telomerase activity, inhibition of metastasis, prevention of circadian disruption, anti-angiogenesis and stimulation of cell differentiation

To date, no treatment modality has demonstrated its clear superiority for leukoplakia. There are many pathways by which melatonin can be used beneficially for management oral leukoplakia.

DETAILED DESCRIPTION:
The World Health Organization (W.H.O). defines oral potentially malignant disorders (OPMDs) as "A histologically proven lesion that is associated with a significantly increased risk of malignant transformation."Oral leukoplakia is the most commonly occurring oral potentially malignant disorder. According to World Health Organisation (WHO), it is defined as "predominantly white plaques of questionable risk having excluded other known diseases or disorders that carry no increased risk for cancer."Leukoplakia has a prevalence rate of 1-4% in the world and 0.2% to 5.2% in Indian Subcontinent, with a malignant transformation rate (MTR) of 0.13% to 10%.

The risk factors include- a) Smokeless and smoking tobacco b) Ultraviolet radiation c) Associated infections like candida, Human papilloma virus (HPV), Epstein Bar Virus (EBV) d) Synergistic effects of alcohol e) Epithelial atrophy due to conditions like syphilis, vitamin deficiencies, iron deficiencies f) trauma.

There are mainly two types of leukoplakia- homogenous and non-homogenous. When widespread or multiple patches of leukoplakia are noted, the term proliferative verrucous leukoplakia (PVL) is used. The homogenous leukoplakias have a lower risk of malignant transformation (0.6%-5%) as compared to non-homogenous (20-25%), while its highest for PVL (61%). The MTR is also high in lesions of size more than 200 mm, tongue and floor of mouth, female patients, old age, severe dysplasia, HPV and candida associated and DNA Aneuploidy.The presence of dysplasia in the lesions of leukoplakia increases the incidence of malignancy by 30 %.

On exposure to carcinogens, tissue cells proliferate and shrink the cytosolic capacity as an adaptation which can be appreciated as hyperplasia of epithelium in histological sections. The persistence of irritant factor leads to cellular degeneration and atrophy, thus further progressing into irreversible cell damages, leading to apoptosis, genetic damages and malignant transformation. There are many studies which suggest the role of reactive oxygen species and reactive nitrogen species in the initiation and progression of carcinogenesis. The generation of oxidative stresses further lead to DNA damage in later stages. Studies are also done which shows decrease in the serum superoxide dismutase, glutathione reductase, glutathione peroxidase and catalase in the patients of leukoplakia.

It is a well-established fact that, oral cancer development is a two-step process which constitutes the emergence of premalignant disorders and their subsequent conversion into cancer. The asymptomatic nature of leukoplakia makes the scenario more difficult as they go unnoticed, leading to their diagnosis only in the stages of malignant conversion. Medical as well as surgical management of cancer causes a deterioration in quality of life of patients due to potentially harmful side effects. Thus, more focus is necessary for chemoprevention of leukoplakia lesions at the premalignant stages thereby preventing its malignant transformation.

The management of leukoplakia includes both conventional as well as surgical modalities. The conventional approaches include Beta Carotene, Lycopene, ascorbic acid, alpha tocopherol, retinoids. But, no significant results are documented on regression rate and prevention of recurrence of the lesions. Other treatment modalities under the experimental trials include extracts of green tea, inhibitors of cyclo-oxygenase 2, epidermal growth factors, peroxisome proliferator. However, there is no generally approved standard systemic therapy so far. Local surgical procedures include photodynamic therapy, laser therapy, cryotherapy and excision.

Melatonin chemically N-acetyl-5-methoxytryptamine is a hormone produced in the pineal gland. It is synthesised from the amino acid, tryptophan. The basic physiological function of melatonin is to control day night cycle and hence is commonly used in insomnia, jet lag and some other psychological disorders.

Melatonin has been proved to exert oncostatic properties through various mechanisms like potent antioxidant effect, antiproliferative functions, stimulation of anticancer immunity, antiangiogenic effects, modulation of oncogene expression and anti-inflammatory. It also exhibits anti candidal and radioprotective effect on the oral mucosa. Thus, melatonin may be helpful in treatment of oral leukoplakia.

Therefore, this study intends to evaluate the effect of topical application of melatonin on clinical response as well as on histopathological and immunohistochemistry findings of leukoplakia.

ELIGIBILITY:
Inclusion Criteria:

Clinically and histologically proven cases of leukoplakia associated with tobacco.

With age 18 years and above. Willing and able to participate in the study and signed informed consent.

Exclusion Criteria:

Patients suspicious of malignant transformation of the lesion with frank ulceration or growth.

Patients consuming or have consumed drugs for treatment of leukoplakia.

Patients who have red or white lesions persisting after radiotherapy treatment

Patients with acquired and congenital immunodeficiency disorders like AIDS, chemotherapy, addiction to injectable opioids and any other significant medical or systemic or autoimmune conditions.

Pregnancy or lactation phase.

Known allergy to melatonin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the size of the lesion. | four and a half months
  measurement of the lesion and scored according to RECIST criteria

SECONDARY OUTCOMES:
Degree of dysplasia | four and a half months
  Grading of dysplasia according to Speight classification (2007).
Expression of immunopositivity of ki67 cells in the lesion. | four and a half months
  Percentage of a total number of Ki-67 positive cells to a total number of cells will be primarily deducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Post graduate institute of dental sciences, Rohtak, Haryana, India